CLINICAL TRIAL: NCT02203136
Title: Improving Clinical Staging for Muscle Invasive Bladder Cancer Through Molecular Profiling and Improved Imaging
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: PA13-0942
Record Dates: First submitted 2014-07-25; First posted 2014-07-29 (Estimated); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Bladder Cancer
Keywords: Bladder cancer; Muscle invasive bladder cancer; MIBC; Biopsy specimen molecular profiling; Bladder surgery; Magnetic resonance imaging; MRI; Trans urethral resection of bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — At the time of biopsy, a portion of the fresh human tumor biopsy samples utilized for DNA and RNA extraction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Muscle Invasive Bladder Cancer (MIBC): During bladder cancer surgery, whole genome gene expression array assays obtained on tumor biopsy specimens. Analysis to determine biologic subtypes which will then be correlated with final pathology, identifying the subtype(s) associated with noc-MIBC. 3 Tesla pelvic magnetic resonance imaging (MRI) performed four weeks after bladder cancer surgery.
  Interventions: Procedure: Tissue Biopsy; Procedure: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Procedure: Tissue Biopsy — During bladder cancer surgery, tissue specimen taken for molecular profiling.
Procedure: Magnetic Resonance Imaging (MRI) — 3 Tesla pelvic magnetic resonance imaging (MRI) performed four weeks after bladder cancer surgery.
  Other Names: MRI

SUMMARY:
The goal of this research study is to improve detection of cancer outside of the bladder through genetic testing and improved imaging.

DETAILED DESCRIPTION:
If participant agrees to take part in the study, a piece of the tumor that is removed during the biopsy will be collected for research purposes. The tissue will be sent to the laboratory for genetic testing.

If they have had a computed tomography scan (CT scan) or magnetic resonance imaging scan (MRI) recently, information collected from the scan will be collected. If they have not had one recently, they will have an MRI with contrast as part of this study. They will receive a separate consent form for this MRI scan.

The results of the test will be given to their doctor, but the results will not be used to decide their treatment.

After they have surgery, information will be collected from their medical records, such as their diagnosis.

Length of Study:

* Their participation on this study will be over once their surgery is completed.
* This is an investigational study.

Up to 100 participants will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with biopsy proven bladder cancer of any age will be eligible for enrollment.

Exclusion Criteria:

1. Contraindication to pelvic MRI (metallic implants/hardware, claustrophobia)
2. Participants who have previously received chemotherapy as part of multimodal therapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants scheduled for bladder cancer surgery and biopsy from the Department of Urology at MD Anderson Cancer Center in Houston, Texas.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2014-06-25 (Actual); Primary Completion 2019-05-16 (Actual); Study Completion 2019-05-16 (Actual)

PRIMARY OUTCOMES:
Detection Improvement of Cancer Outside of the Bladder | 4 weeks
  Improved cross sectional imaging with pelvic MRI, and biopsy specimen molecular profiling used to identify muscle invasive bladder cancer (noc-MIBC). Analysis to determine biologic subtypes which will then be correlated with final pathology, identifying the subtype(s) associated with noc-MIBC.

CONTACTS AND LOCATIONS:
Overall Officials: Neema Navai, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org